CLINICAL TRIAL: NCT02528435
Title: Role of Pharmacogenetic and Psychological Factors in Methotrexate Tolerance: Studies in Children With Chronic Arthritis and Children With Leukemia
Brief Title: Understanding Methotrexate Induced Gastrointestinal Intolerance in Juvenile Idiopathic Arthritis and Childhood Leukemia
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: MTX Project
Record Dates: First submitted 2015-05-28; First posted 2015-08-19 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2017-04

CONDITIONS: Juvenile Idiopathic Arthritis; ALL
Keywords: Methotrexate
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample to SNP analysis - see project description
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- JIA patients: observationational study including children diagnosed with JIA. Patients aged 9 years and above, whom are treated with low-dose MTX may be included.
- ALL patients: observationational study including children diagnosed with ALL. Patients aged 9 years and above, whom are in maintenance treatment with low-dose MTX may be included.

SUMMARY:
Methotrexate is a cornerstone in the treatment of childhood leukemia. When given in high-dose as part of the initial phase of treatment, gastrointestinal toxicity is a known problem. However when children reach maintenance treatment with low-dose methotrexate this is not described as a significant challenge. Children with juvenile idiopathic arthritis are another patient group receiving low-dose methotrexate. Among these patients gastrointestinal intolerance is such a significant problem that treatment may be ceased. The aim of this project is to create a greater understanding of gastrointestinal intolerance associated to low-dose methotrexate treatment by investigating the differences between these two patient groups, investigating genetic and psychological factors.

DETAILED DESCRIPTION:
Background:

Childhood leukemia (Acute Lymphoblastic Leukemia, ALL) is the most frequent malignancy in the pediatric population (1). Survival rates have reached above 85% due to advances in chemotherapy. High-dose methotrexate (MTX) is a mainstay in the treatment of ALL (2-4). Gastrointestinal toxicity is a well known challenge associated to high-dose MTX treatment (5). However this is not described as a significant problem among these children when they reach maintenance treatment and receive low-dose MTX treatment. Children with Juvenile Idiopathic Arthritis (JIA) also receive low-dose MTX treatment. Among these patients MTX induced gastrointestinal intolerance is a significant problem. Studies have shown that more than half of the JIA patients have problems tolerating MTX because of nausea which may lead to cessation of treatment (6,7). It is largely unknown why MTX causes nausea but both pharmacogenetic and psychological factors are thought to play a role (8).

JIA is the most common chronic pediatric rheumatic disease. Without treatment the disease causes significant short- and long-term disability and quality of life impairment. Prognosis has greatly improved within recent years as a result of substantial progress in disease management and MTX is a mainstay in the treatment of JIA (9-13).

The aim of this project is to create a greater understanding of MTX induced gastrointestinal intolerance among children with leukemia and children with JIA. The project will focus on nausea and investigate the level of nausea in the two patient groups and compare if a difference does exist. The investigators will further investigate pharmacogenetic and psychological factors and their relation to the patients' level of nausea.

Pharmacogenetic background:

MTX is absorbed from the gastrointestinal tract and transported to the bloodstream by transporter proteins in the enterocytes. Elimination of MTX is primarily renal but a percentage of MTX passes through enterohepatic circulation first (14,15). Studies on the use of high-dose MTX treatment to children with ALL suggest that fast hepatic clearance of MTX increases the degree of gastrointestinal toxicity. It has further been shown that patients with mutations (Single Nucleotide Peptides, SNPs) in the gene encoding the hepatic transporter protein SLCO1B1, responsible for transporting MTX into the liver, have less gastrointestinal toxicity to high-dose MTX (16). The transporter protein encoded by SLC19A1 is placed both in the liver and the enterocytes (15).

Studies on adult patients diagnosed with either psoriasis or rheumatoid arthritis and treated with low-dose MTX, and studies on ALL patients in high-dose MTX show that SLC19A1 is associated to the concentration of MTX in plasma and erythrocytes as well as MTX-related toxicity (1,17-20). Transporter proteins that transport MTX out of the liver and into the bile ducts are encoded by ABCC2 and ABCB1(15). Studies on adult patients with rheumatoid arthritis in low-dose MTX, adults with Chronic Myeloid Leukemia and studies on ALL patients in high-dose MTX have shown that both genes are pharmacokinetically important and ABCC2 has further been shown associated to MTX-related gastrointestinal toxicity (5,21-24). Previous studies on patients with rheumatoid arthritis, childhood leukemia and JIA have shown that the frequency of clinically relevant SNPs in genes encoding MTX-related transporter proteins are: SLCO1B1 (70.3%), ABCB1 (20.6%), ABCC2 (56.8%), SLC19A1 (31%) (5,16,17,19,21,25-28).The investigators therefore believe it conceivable to find the selected genetic polymorphisms for MTX-related transporter proteins in the participating study population.

Pharmocogenetic Aims:

Investigate if MTX-related gastrointestinal intolerance is associated to the enterohepatic circulation. Specifically, to determine if SNPs in genes encoding MTX-related liver transporter proteins are associated to the level of drug induced gastrointestinal side effects.

Pharmacogenetic Hypotheses:

Patients with SNPs in genes encoding MTX-related transporter proteins in the liver have a lower level of enterohepatic circulation of MTX and thus have a lower level of nausea than other patients.

Psychological Background:

Studies on adult cancer patients have shown that psychologically based nausea occurring after treatment with chemotherapy is a possible explanation for the nausea which is out of proportion with the medicine's emetogenic potential. It is also a possible explanation for the great variation in the level of cancer patients' nausea after the same type of chemotherapy (29,30). Studies on children in chemotherapy for different cancers have shown that psychological factors, such as coping strategies and anxiety, affect the degree of chemotherapy associated nausea and vomiting (31-33). The investigators want to investigate if this is also the case for children with leukemia in maintenance treatment with low-dose MTX as well as JIA patients in low-dose MTX-treatment.

Psychological aims:

To investigate if the nausea-coping strategies and anxiety level of the study population are associated to the degree of MTX-induced gastrointestinal intolerance. And investigate if there is a difference between the two patient groups.

Psychological hypotheses:

Insufficient psychological coping strategies and high level of anxiety may cause psychologically based nausea. Thus patients with a high level of anxiety and insufficient coping strategies will have a higher degree of nausea to MTX treatment than other patients.

Perspectives This project will contribute to a greater understanding of MTX-induced intolerance in children with leukemia and JIA. This will also be beneficial for all other children who receive low-dose MTX treatment. The project will optimize the maintenance treatment of childhood leukemia and the treatment of JIA by using patient SNP genotypes to determine who can tolerate MTX and who cannot. Additionally, identify patients where psychological intervention may diminish MTX-induced nausea.

Materials and methods

The study population comprises:

1. Children diagnosed with ALL in maintenance treatment
2. Children diagnosed with JIA according to ILAR criteria

For inclusion/exclusion criteria see under "Eligibility Criteria". For each patient a list of disease specific characteristics will be noted. The level of MTX-induced intolerance is determined by an electronic "nausea-diary" for four weeks, containing a "faces of nausea scale" based on a "faces of pain scale" (34). The gastrointestinal side effects will further be evaluated by a Methotrexate-Intolerance-Severity-Score questionnaire (MISS) (35).

Pharmacogenetic methods:

Blood samples on each patient will be used to determine the prevalence of SNPs in genes encoding MTX-related transporter proteins (genes including: SLCO1B1, SLC19A1, ABCC2, ABCB1). The genetic analysis will be performed at the Institute of Biomedicine, Aarhus University. Genotyping are carried out using the Sequenom MassARRAY Genotyping system (Sequenom, San Diego, CA). In brief multiplex PCR are performed in 5 μl reactions containing 10 ng of genomic DNA, 1.25 x PCR buffer, 0.5 mM dNTP, 100nM of each primer and 0.5U Taq polymerase using standard cycling conditions. The PCR products are then treated with SAP and the probe extension reaction (iPLEX) carried according to the iPLEX standard protocol (Sequenom). The desalted samples are analyzed using a Bruker matrix assisted laser desorption/ionization-time of flight (MALDI-TOF) mass spectrometer (Sequenom) and the genotypes determined using the MassARRAY Typer 3.4 software (Sequenom). The blood sample will also be used to measure the concentration of MTX-polyglutamates in the erythrocytes (Ery-MTX-PG). The measurement of Ery-MTX-PG will be performed by HPLC-technique at the children's oncology lab, Rigshospitalet, Copenhagen, Denmark.

2) Psychological methods: The patients' coping strategies will be investigated using a nausea-coping-questionnaire developed from a pain-coping questionnaire, which has specifically been developed for children and previously been translated to Danish, validated and used in earlier studies. It consists of eight subscales of main coping strategies: Information seeking, problem solving, seeking social support, positive self-statements, behavioral distraction, cognitive distraction, externalizing and internalizing/catastrophizing (36,37,39,40). The patients' level of anxiety will be assessed by "Beck Youth Inventories" (BYI), which previously have been translated into Danish and validated. The BYI is brief and easy to use. It consists of 20 sentences that investigate fear, worrying and physiological symptoms associated with anxiety (38).

Statistics Power calculation: This is based on the primary target measure (the degree of nausea) quantified by the "faces of nausea scale" in the nausea diary. The scale has the end points: "no nausea" and "extreme nausea", in numbers 0 to 5. Results from an earlier study using the faces of pain scale show that mean scores were 0.74 (SD=0.70) and 0.91(SD=0.86) (36). From a clinical assessment the investigators expect the mean nausea score for the group of JIA patients to be 2.5 and 1 for the ALL patients. The standard deviation is expected to be similar to the study above (SD=0.9). If the level of significance (alpha) is 0.05, the power is 80% and the ratio between the group sizes is 2, then the calculated size of the study population will be 10 patients in the JIA group and 5 in the ALL group. If the mean nausea score only is 2 for the group of JIA patients, but still 1 for the group of ALL patients, and the standard deviation is greater than expected, SD=2. But alpha still is 0.05, the power is 80%, and the ratio between the group sizes is still 2. Then the calculated size of the study population will be 96 patients in the JIA group and 48 in the ALL group.

Research Plan

The research group consists of:

From Department of Pediatrics, Aarhus University Hospital Skejby:

Main applicant: Nini Kyvsgaard Brix Nørgaard, PhD-student (enrolled at Aarhus University), M.D.

Main supervisor: Troels Herlin, Professor, DMSc; Co-supervisor: Torben Stamm Mikkelsen, MD, PhD.

From Institute of Biomedicine, Aarhus University:

Co-supervisor: Thomas Juhl Corydon, Associate Professor, PhD, Deputy Head of Institute for Biomedicine, Aarhus University.

From Institute for Psychology, Aarhus University:

Co-Supervisor: Mikael Thastum, Professor, PhD, Head of Clinical Psychology, Aarhus University.

The PhD-student will perform and coordinate the daily execution of the project with guidance from the group of supervisors. The first and second year of the project will be dedicated to the collection of patient data and blood samples. Firstly, the inclusion of the JIA patients will commence. Then the inclusion of the ALL patients. The third year will be dedicated to analysis of gene polymorphisms and MTX levels, data analysis and compilation of manuscripts for publication. The research group has extensive research experience and clinical expertise within this area.

Feasibility The laboratory facilities to take the blood samples and carry out the initial handling of them are available. The final analysis will be performed as specified under 'pharmacogenetic methods'. The investigators have access to software to perform the questionnaires electronically, as well as access to statistical support.

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed with JIA according to ILAR criteria, whom are followed at the departments of pediatrics at Aarhus University Hospital Skejby and Odense University Hospital.
* and children diagnosed with ALL, whom are followed at the departments of pediatrics at Aarhus University Hospital Skejby, Aalborg University Hospital, Odense University Hospital and Rigshospitalet.
* aged 9 years and above
* currently treated with low-dose MTX for at least six weeks

Exclusion Criteria:

* Children with cognitive difficulties will be excluded
* Children without ability to speak Danish will be excluded.

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: see under project - and group description
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Methotrexate-induced Nausea | after project year 2 there will be final data analysis
  "faces nausea scale" in the nausea diary

SECONDARY OUTCOMES:
Methotrexate Intolerance | after project year 2 there will be final data analysis
  Methotrexate Intolerance Severity Score by Bulatovic et al (see citation list)

REFERENCES:
- [Background] Laverdiere C, Chiasson S, Costea I, Moghrabi A, Krajinovic M. Polymorphism G80A in the reduced folate carrier gene and its relationship to methotrexate plasma levels and outcome of childhood acute lymphoblastic leukemia. Blood. 2002 Nov 15;100(10):3832-4. doi: 10.1182/blood.V100.10.3832. PMID 12411325
- [Background] Levinsen M, Rosthoj S, Nygaard U, Heldrup J, Harila-Saari A, Jonsson OG, Bechensteen AG, Abrahamsson J, Lausen B, Frandsen TL, Weinshilboum RM, Schmiegelow K. Myelotoxicity after high-dose methotrexate in childhood acute leukemia is influenced by 6-mercaptopurine dosing but not by intermediate thiopurine methyltransferase activity. Cancer Chemother Pharmacol. 2015 Jan;75(1):59-66. doi: 10.1007/s00280-014-2613-7. Epub 2014 Oct 28. PMID 25347948
- [Background] Lopez-Lopez E, Gutierrez-Camino A, Bilbao-Aldaiturriaga N, Pombar-Gomez M, Martin-Guerrero I, Garcia-Orad A. Pharmacogenetics of childhood acute lymphoblastic leukemia. Pharmacogenomics. 2014 Jul;15(10):1383-98. doi: 10.2217/pgs.14.106. PMID 25155938
- [Background] Pui CH, Schrappe M, Ribeiro RC, Niemeyer CM. Childhood and adolescent lymphoid and myeloid leukemia. Hematology Am Soc Hematol Educ Program. 2004:118-45. doi: 10.1182/asheducation-2004.1.118. PMID 15561680
- [Background] Rau T, Erney B, Gores R, Eschenhagen T, Beck J, Langer T. High-dose methotrexate in pediatric acute lymphoblastic leukemia: impact of ABCC2 polymorphisms on plasma concentrations. Clin Pharmacol Ther. 2006 Nov;80(5):468-76. doi: 10.1016/j.clpt.2006.08.012. PMID 17112803
- [Background] Gutierrez-Suarez R, Burgos-Vargas R. The use of methotrexate in children with rheumatic diseases. Clin Exp Rheumatol. 2010 Sep-Oct;28(5 Suppl 61):S122-7. Epub 2010 Oct 28. PMID 21044445
- [Background] Wallace CA. The use of methotrexate in childhood rheumatic diseases. Arthritis Rheum. 1998 Mar;41(3):381-91. doi: 10.1002/1529-0131(199803)41:33.0.CO;2-3. No abstract available. PMID 9506564
- [Background] Moncrieffe H, Hinks A, Ursu S, Kassoumeri L, Etheridge A, Hubank M, Martin P, Weiler T, Glass DN, Thompson SD, Thomson W, Wedderburn LR. Generation of novel pharmacogenomic candidates in response to methotrexate in juvenile idiopathic arthritis: correlation between gene expression and genotype. Pharmacogenet Genomics. 2010 Nov;20(11):665-76. doi: 10.1097/FPC.0b013e32833f2cd0. PMID 20827233
- [Background] Nordal E, Zak M, Aalto K, Berntson L, Fasth A, Herlin T, Lahdenne P, Nielsen S, Straume B, Rygg M; Nordic Study Group of Pediatric Rheumatology. Ongoing disease activity and changing categories in a long-term nordic cohort study of juvenile idiopathic arthritis. Arthritis Rheum. 2011 Sep;63(9):2809-18. doi: 10.1002/art.30426. PMID 21560116
- [Background] Giannini EH, Ilowite NT, Lovell DJ, Wallace CA, Rabinovich CE, Reiff A, Higgins G, Gottlieb B, Singer NG, Chon Y, Lin SL, Baumgartner SW; Pediatric Rheumatology Collaborative Study Group. Long-term safety and effectiveness of etanercept in children with selected categories of juvenile idiopathic arthritis. Arthritis Rheum. 2009 Sep;60(9):2794-804. doi: 10.1002/art.24777. PMID 19714630
- [Background] Beresford MW, Baildam EM. New advances in the management of juvenile idiopathic arthritis--1: non-biological therapy. Arch Dis Child Educ Pract Ed. 2009 Oct;94(5):144-50. doi: 10.1136/adc.2008.144576. PMID 19770494
- [Background] Hashkes PJ, Laxer RM. Medical treatment of juvenile idiopathic arthritis. JAMA. 2005 Oct 5;294(13):1671-84. doi: 10.1001/jama.294.13.1671. PMID 16204667
- [Background] Salliot C, van der Heijde D. Long-term safety of methotrexate monotherapy in patients with rheumatoid arthritis: a systematic literature research. Ann Rheum Dis. 2009 Jul;68(7):1100-4. doi: 10.1136/ard.2008.093690. Epub 2008 Dec 5. PMID 19060002
- [Background] Steinberg SE, Campbell CL, Bleyer WA, Hillman RS. Enterohepatic circulation of methotrexate in rats in vivo. Cancer Res. 1982 Apr;42(4):1279-82. PMID 7060005
- [Background] Mikkelsen TS, Thorn CF, Yang JJ, Ulrich CM, French D, Zaza G, Dunnenberger HM, Marsh S, McLeod HL, Giacomini K, Becker ML, Gaedigk R, Leeder JS, Kager L, Relling MV, Evans W, Klein TE, Altman RB. PharmGKB summary: methotrexate pathway. Pharmacogenet Genomics. 2011 Oct;21(10):679-86. doi: 10.1097/FPC.0b013e328343dd93. No abstract available. PMID 21317831
- [Background] Trevino LR, Shimasaki N, Yang W, Panetta JC, Cheng C, Pei D, Chan D, Sparreboom A, Giacomini KM, Pui CH, Evans WE, Relling MV. Germline genetic variation in an organic anion transporter polypeptide associated with methotrexate pharmacokinetics and clinical effects. J Clin Oncol. 2009 Dec 10;27(35):5972-8. doi: 10.1200/JCO.2008.20.4156. Epub 2009 Nov 9. PMID 19901119
- [Background] Gregers J, Christensen IJ, Dalhoff K, Lausen B, Schroeder H, Rosthoej S, Carlsen N, Schmiegelow K, Peterson C. The association of reduced folate carrier 80G>A polymorphism to outcome in childhood acute lymphoblastic leukemia interacts with chromosome 21 copy number. Blood. 2010 Jun 10;115(23):4671-7. doi: 10.1182/blood-2010-01-256958. Epub 2010 Mar 24. PMID 20335220
- [Background] Kishi S, Cheng C, French D, Pei D, Das S, Cook EH, Hijiya N, Rizzari C, Rosner GL, Frudakis T, Pui CH, Evans WE, Relling MV. Ancestry and pharmacogenetics of antileukemic drug toxicity. Blood. 2007 May 15;109(10):4151-7. doi: 10.1182/blood-2006-10-054528. Epub 2007 Jan 30. PMID 17264302
- [Background] Dervieux T, Kremer J, Lein DO, Capps R, Barham R, Meyer G, Smith K, Caldwell J, Furst DE. Contribution of common polymorphisms in reduced folate carrier and gamma-glutamylhydrolase to methotrexate polyglutamate levels in patients with rheumatoid arthritis. Pharmacogenetics. 2004 Nov;14(11):733-9. doi: 10.1097/00008571-200411000-00004. PMID 15564880
- [Background] Campalani E, Arenas M, Marinaki AM, Lewis CM, Barker JN, Smith CH. Polymorphisms in folate, pyrimidine, and purine metabolism are associated with efficacy and toxicity of methotrexate in psoriasis. J Invest Dermatol. 2007 Aug;127(8):1860-7. doi: 10.1038/sj.jid.5700808. Epub 2007 Apr 5. PMID 17410198
- [Background] Yamakawa Y, Hamada A, Nakashima R, Yuki M, Hirayama C, Kawaguchi T, Saito H. Association of genetic polymorphisms in the influx transporter SLCO1B3 and the efflux transporter ABCB1 with imatinib pharmacokinetics in patients with chronic myeloid leukemia. Ther Drug Monit. 2011 Apr;33(2):244-50. doi: 10.1097/FTD.0b013e31820beb02. PMID 21311410
- [Background] Ranganathan P, Culverhouse R, Marsh S, Mody A, Scott-Horton TJ, Brasington R, Joseph A, Reddy V, Eisen S, McLeod HL. Methotrexate (MTX) pathway gene polymorphisms and their effects on MTX toxicity in Caucasian and African American patients with rheumatoid arthritis. J Rheumatol. 2008 Apr;35(4):572-9. Epub 2008 Mar 15. PMID 18381794
- [Background] Stamp LK, O'Donnell JL, Chapman PT, Zhang M, James J, Frampton C, Barclay ML. Methotrexate polyglutamate concentrations are not associated with disease control in rheumatoid arthritis patients receiving long-term methotrexate therapy. Arthritis Rheum. 2010 Feb;62(2):359-68. doi: 10.1002/art.27201. PMID 20112376
- [Background] Stamp LK, Chapman PT, O'Donnell JL, Zhang M, James J, Frampton C, Barclay ML, Kennedy MA, Roberts RL. Polymorphisms within the folate pathway predict folate concentrations but are not associated with disease activity in rheumatoid arthritis patients on methotrexate. Pharmacogenet Genomics. 2010 Jun;20(6):367-76. doi: 10.1097/FPC.0b013e3283398a71. PMID 20386493
- [Background] Wessels JA, de Vries-Bouwstra JK, Heijmans BT, Slagboom PE, Goekoop-Ruiterman YP, Allaart CF, Kerstens PJ, van Zeben D, Breedveld FC, Dijkmans BA, Huizinga TW, Guchelaar HJ. Efficacy and toxicity of methotrexate in early rheumatoid arthritis are associated with single-nucleotide polymorphisms in genes coding for folate pathway enzymes. Arthritis Rheum. 2006 Apr;54(4):1087-95. doi: 10.1002/art.21726. PMID 16572443
- [Background] van Ede AE, Laan RF, Blom HJ, Huizinga TW, Haagsma CJ, Giesendorf BA, de Boo TM, van de Putte LB. The C677T mutation in the methylenetetrahydrofolate reductase gene: a genetic risk factor for methotrexate-related elevation of liver enzymes in rheumatoid arthritis patients. Arthritis Rheum. 2001 Nov;44(11):2525-30. doi: 10.1002/1529-0131(200111)44:113.0.co;2-b. PMID 11710708
- [Background] Schmeling H, Biber D, Heins S, Horneff G. Influence of methylenetetrahydrofolate reductase polymorphisms on efficacy and toxicity of methotrexate in patients with juvenile idiopathic arthritis. J Rheumatol. 2005 Sep;32(9):1832-6. PMID 16142884
- [Background] Dervieux T, Furst D, Lein DO, Capps R, Smith K, Walsh M, Kremer J. Polyglutamation of methotrexate with common polymorphisms in reduced folate carrier, aminoimidazole carboxamide ribonucleotide transformylase, and thymidylate synthase are associated with methotrexate effects in rheumatoid arthritis. Arthritis Rheum. 2004 Sep;50(9):2766-74. doi: 10.1002/art.20460. PMID 15457444
- [Background] Watson M, McCarron J, Law M. Anticipatory nausea and emesis, and psychological morbidity: assessment of prevalence among out-patients on mild to moderate chemotherapy regimens. Br J Cancer. 1992 Nov;66(5):862-6. doi: 10.1038/bjc.1992.374. PMID 1419628
- [Background] Watson M, Meyer L, Thomson A, Osofsky S. Psychological factors predicting nausea and vomiting in breast cancer patients on chemotherapy. Eur J Cancer. 1998 May;34(6):831-7. doi: 10.1016/s0959-8049(97)10146-0. PMID 9797694
- [Background] Tyc VL, Mulhern RK, Fairclough D, Ward PM, Relling MV, Longmire W. Chemotherapy induced nausea and emesis in pediatric cancer patients: external validity of child and parent emesis ratings. J Dev Behav Pediatr. 1993 Aug;14(4):236-41. PMID 8408666
- [Background] Tyc VL, Mulhern RK, Jayawardene D, Fairclough D. Chemotherapy-induced nausea and emesis in pediatric cancer patients: an analysis of coping strategies. J Pain Symptom Manage. 1995 Jul;10(5):338-47. doi: 10.1016/0885-3924(95)00019-u. PMID 7673766
- [Background] Dolgin MJ, Katz ER. Conditioned aversions in pediatric cancer patients receiving chemotherapy. J Dev Behav Pediatr. 1988 Apr;9(2):82-5. PMID 3366914
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Bulatovic M, Heijstek MW, Verkaaik M, van Dijkhuizen EH, Armbrust W, Hoppenreijs EP, Kamphuis S, Kuis W, Egberts TC, Sinnema G, Rademaker CM, Wulffraat NM. High prevalence of methotrexate intolerance in juvenile idiopathic arthritis: development and validation of a methotrexate intolerance severity score. Arthritis Rheum. 2011 Jul;63(7):2007-13. doi: 10.1002/art.30367. PMID 21437879
- [Background] Thastum M, Herlin T. Pain-specific beliefs and pain experience in children with juvenile idiopathic arthritis: a longitudinal study. J Rheumatol. 2011 Jan;38(1):155-60. doi: 10.3899/jrheum.091375. Epub 2010 Oct 15. PMID 20952477
- [Background] Thastum M, Herlin T, Zachariae R. Relationship of pain-coping strategies and pain-specific beliefs to pain experience in children with juvenile idiopathic arthritis. Arthritis Rheum. 2005 Apr 15;53(2):178-84. doi: 10.1002/art.21081. PMID 15818646
- [Background] Thastum M, Ravn K, Sommer S, Trillingsgaard A. Reliability, validity and normative data for the Danish Beck Youth Inventories. Scand J Psychol. 2009 Feb;50(1):47-54. doi: 10.1111/j.1467-9450.2008.00690.x. Epub 2008 Oct 22. PMID 18980602
- [Background] Thastum M, Zachariae R, Herlin T. Pain experience and pain coping strategies in children with juvenile idiopathic arthritis. J Rheumatol. 2001 May;28(5):1091-8. PMID 11361195
- [Background] Thastum M, Zachariae R, Scholer M, Herlin T. A Danish adaptation of the Pain Coping Questionnaire for children: preliminary data concerning reliability and validity. Acta Paediatr. 1999 Feb;88(2):132-8. doi: 10.1080/08035259950170277. PMID 10102143